CLINICAL TRIAL: NCT01761630
Title: ALXR/FPR Mediated Signaling in Severe Asthma (AMSA)-The Severe Asthma Research Program (SARP) III
Brief Title: The Severe Asthma Research Program III-Boston Clinical Site
Acronym: SARPIII-AMSA
Status: Completed | Type: Observational
Sponsor: Elliot Israel, MD (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Elliot Israel, MD, Professor of Medicine, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Other Study IDs: 2012P001528
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Asthma
Keywords: Asthma; Severe Asthma; SARP
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CBC/Diff, Total IgE, Serum, Plasma, DNA, RNA Urine EBC Sputum: Supernatant, Cell Pellet Bronch: BAl, Bronchial Brushings, Bronchial Biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Severe Asthma: We will classify subjects as having severe asthma using the following stages:
  Stage 1: Subjects must have asthma which requires treatment with high-dose inhaled corticosteroids plus a 2nd controller, or systemic corticosteroids with or without a 2nd controller to prevent it from becoming uncontrolled or which remains uncontrolled despite this therapy
  Stage 2: Assess for uncontrolled asthma by any one of the following criteria:
  1. Poor symptom control evidenced by an Asthma Control Questionnaire score consistently > 1.5 or an Asthma Control Test Score < 20 or not well controlled by NAEPP or GINA asthma treatment guidelines
  2. Frequent severe exacerbations as reflected by ≥ 2 bursts of systemic corticosteroids (> 3 days each) in the previous 12 months
  3. Serious exacerbations reflected by at least one hospitalization, ICU stay or mechanical ventilation in the previous 12 months
  4. Presence of airflow limitation evidenced by FEV1 < 80% predicted (in the face of reduced FEV1/FVC)
- Non-severe Asthma: Those with mild-to-moderate persistent asthma as defined by the NAEPP EPR-3 guidelines.
- Healthy Control: The purpose of the SARP Control Sub-study is to generate reference data for outcomes measured in biospecimens collected from asthmatic subjects enrolled in the SARP Longitudinal Protocol.
  Seven healthy subjects between the ages of 18-65 will be enrolled.

SUMMARY:
Asthma is a disease characterized by inflammation in the airways. The body naturally makes compounds that reduce inflammation. Unfortunately, for patients with severe asthma, the pathway these compounds use to reduce inflammation seems to be perturbed. Investigators have chosen to focus on the anti-inflammatory compounds called lipoxins and how they work through the "ALX Axis", a name given to the ALX receptor pathway and its ligands. Work from the Brigham and Women's Hospital has suggested that in patients with severe asthma, the ALX axis may not work properly and therefore may not shut off inflammation as expected. Also, there is information to suggest that in some cases, steroids (prednisone and similar drugs), which are commonly used to treat asthma, may affect the ALX axis in a negative way, paradoxically making the inflammation worse instead of better.

As part of the NIH Severe Asthma Research Program the Asthma Research Center's goal is to identify what causes the problems in the ALX axis in severe asthma. To do so, participants with severe asthma will be compared to participants with milder forms of asthma. Investigators will use samples taken directly from the lungs of people with asthma, as well as blood, urine and CT scans of the lungs to better understand how the ALX axis changes both before and after corticosteroid treatment and throughout a three year span. Participants will come into the Asthma Research Center to have the procedures done.

Investigators expect participants will perform breathing tests and complete questionnaires and diaries. To better understand if corticosteroids negatively affect the ALX axis in severe asthma, researchers will take samples before and after a one time steroid injection equivalent to a prednisone treatment for asthma. Participants will perform two bronchoscopy procedures, before and after corticosteroid treatment, where biopsies and cells will be obtained from the participant's lungs. Investigators will use these samples to observe any changes that the corticosteroid may have on the ALX axis. At the end of the study, researchers at the Brigham and Women's Hospital expect to understand the ALX axis in such a way that will allow them to formulate new therapies and drug targets to treat people with asthma, especially severe asthma, more effectively.

In Boston, this study will be run together by the Asthma Research Center at the Brigham and Women's Hospital (adults) and Boston Children's Hospital (children).

DETAILED DESCRIPTION:
Severe asthma accounts for the majority of the morbidity and mortality related to asthma. It is characterized by persistent airway inflammation despite anti-inflammatory therapy, persistent airway hyperresponsiveness, and "remodeling" of the airways that includes fibrosis. Lipoxin A4 (LXA4) and 15-epimer-LXA4 are lipid-derived mediators that have been shown to promote anti-inflammatory and pro-resolving cellular responses through their effects at ALX/FPR2 receptors. They promote resolution of inflammation, inhibit airway hyperresponsiveness, and counteract pro-fibrotic processes. Investigators at the Brigham and Women's Hospital and others have shown that the ALX effector pathway and its constituent ligands (ALX axis) is perturbed in severe asthma (SA) compared with non-severe asthma (NSA). Specifically, in SA LXA4 production is decreased and ALX/FPR2 receptor expression is reduced. Further, investigators at the Brigham and Women's Hospital have shown that low levels of lipoxins, relative to pro phlogistic leukotrienes, are associated with reduced airway function (FEV1). Considering these data and the function of the ALX axis, it appears that perturbations of constituents of this axis could identify, and perhaps underlie, several of the processes that characterize severe, progressive asthma. Further to this point, work in progress being done at the Brigham and Women's Hospital indicates that corticosteroids (CS) interactions with the ALX axis may underlie some of these perturbations. CS can decrease the production of LXA4. More importantly, while CS increase production of pro-resolving annexin A1, they also appear to promote pro-inflammatory signaling through ALX/FPR2 via upregulation of serum amyloid A (SAA). SAA is expressed in the lung and is associated with exacerbations of COPD.

Hypotheses:

Peripheral blood leukocytes and bronchoalveolar lavage fluids will be obtained from SA and NSA subjects before and after intramuscular triamcinolone at baseline to test the hypothesis that in vivo corticosteroids will reduce pro-inflammatory cellular responses and enhance LXA4-mediated anti-inflammatory responses in the majority of asthmatic subjects. There is a sub-group of individuals with severe asthma in which in vivo corticosteroids will paradoxically increase pro-inflammatory responses. Investigators will also test the hypothesis that such paradoxical signaling can be overcome by lipoxins. In addition, investigators will test the hypothesis that basal p anti-inflammatory responses are dampened in severe asthma.

Investigators at the Brigham and Women's Hospital hypothesize that a cohort of severe asthmatic subjects with impaired counter-regulatory signaling will have a specific ALX axis phenotype that will predispose them to increased inflammation, asthma exacerbations and disease progression.

Investigators will test the hypothesis that in vivo corticosteroids will not increase (and may decrease) LXA4 or 15-epi-LXA4 but will increase annexin A1 and serum amyloid A and that the levels of these compounds post-CS will differ by disease severity, remaining stable over a 3 year interval.

Samples will be obtained at study entry before and after intramuscular triamcinolone to test the hypothesis that in vivo corticosteroids increase ALX/FPR2 expression in leukocytes and airway cells.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6-60
* FEV1 bronchodilator reversibility ≥12% or methacholine PC20 ≤16 mg/mL
* Ability to provide informed consent
* Ability to perform pulmonary function tests

Exclusion Criteria:

* Pregnancy (if undergoing methacholine challenge or bronchoscopy)
* Current smoking
* Smoking history > 10 pack years if ≥ 30 years of age or smoking history > 5 pack years if < 30 years of age (Note: If a subject has a smoking history, no smoking within the past year)
* Other chronic pulmonary disorders associated with asthma-like symptoms, including (but not limited to) cystic fibrosis, chronic obstructive pulmonary disease, chronic bronchitis, vocal cord dysfunction that is the sole cause of asthma symptoms, severe scoliosis or chest wall deformities that affect lung function, or congenital disorders of the lungs or airways
* Participants who cannot undergo bronchoscopy due to: 1) hospitalization for asthma within the 6 weeks prior to bronchoscopy, 2) > 12 asthma exacerbations within the 6 months prior to bronchoscopy, 3) intubation for asthma within the 6 months prior to bronchoscopy, 4) older than 60 years of age, 5) increased corticosteroid use in the 14 days prior to bronchoscopy. (Increased corticosteroid use recognized as a dose which is both numerically at least twice that of baseline, and which is at least 20 mg/day greater than the baseline dose.)
* History of premature birth before 35 weeks gestation
* Planning to relocate from the clinical center area before study completion
* Currently participating in an investigational drug trial
* Unwillingness to receive an intramuscular triamcinolone acetonide injection.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The target recruitment goal for our center is 75% adults (age 18 to 60) and 25% children age 6-17 years. Within the pediatric age group, an attempt will be made to enroll equal numbers of children 6-11 and 12-17 years of age. Similarly, an attempt will be made to enroll at least 50% females and 30% minorities.
  Given the mission of SARP, a diverse sample of subjects with asthma is needed to gain better understanding of asthma and its endotypes. Because there are a number of respiratory disorders that may be confused with asthma or confound asthma assessment, SARP enrollees must meet the all of the eligibility criteria described.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2012-12; Primary Completion 2020-03-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Longitudinal change in maximum bronchodilator (BD) FEV1 response. | Evaluated at Visits 1, 3, 4, 5, 6 (Months 0, 1, 12, 24, 36)
Changes in values of ALX axis ligands and ALX/FPR2 receptor expression before and after corticosteroid treatment in severe asthmatics and non-severe asthmatics. | Evaluated at Visit 2, 2b, 3, 3b (Days 7, 9, 23,25)
  Sputum, blood, and bronchoscopic specimens will be obtained before and after parenteral triamcinolone to directly assess the ALX axis in the airway. Particular attention will be paid to the change in LXA4, 15-epi-LXA4, SAA, and ANXA1 ligands.
Change in CT measures of airway wall thickness (WA%) over 3 years | Evaluated at Visits 2, 6 (Months 0, 36)
  Data will only be collected from adult participants.
Number of severe asthma exacerbations per subject | Evaluated at Visits 1, 2, 3, 3a, 4, 4a, 5, 5a, 6 (Months 0, 1, 2, 6, 12, 18, 24, 30, 36)
Plasma LXA4/CysLT levels and their ability to predict increases or decreases in FEV1, exacerbations, and WA% over time. | Evaluated at Visits 2, 3, 4, 5, 6 (Months 0, 1, 12, 24, 36)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Israel, M.D., Principal Investigator — Brigham and Women's Hospital/Harvard Medical School; Bruce Levy, M.D., Principal Investigator — Brigham and Women's Hospital/Harvard Medical School
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Huang BK, Elicker BM, Henry TS, Kallianos KG, Hahn LD, Tang M, Heng F, McCulloch CE, Bhakta NR, Majumdar S, Choi J, Denlinger LC, Fain SB, Hastie AT, Hoffman EA, Israel E, Jarjour NN, Levy BD, Mauger DT, Sumino K, Wenzel SE, Castro M, Woodruff PG, Fahy JV, Sarp FTNSARP. Persistent mucus plugs in proximal airways are consequential for airflow limitation in asthma. JCI Insight. 2024 Feb 8;9(3):e174124. doi: 10.1172/jci.insight.174124. PMID 38127464
- [Derived] Ash SY, Sanchez-Ferrero GV, Schiebler ML, Rahaghi FN, Rai A, Come CE, Ross JC, Colon AG, Cardet JC, Bleecker ER, Castro M, Fahy JV, Fain SB, Gaston BM, Hoffman EA, Jarjour NN, Lempel JK, Mauger DT, Tattersall MC, Wenzel SE, Levy BD, Washko GR, Israel E, San Jose Estepar R; SARP Investigators. Estimated Ventricular Size, Asthma Severity, and Exacerbations: The Severe Asthma Research Program III Cohort. Chest. 2020 Feb;157(2):258-267. doi: 10.1016/j.chest.2019.08.2185. Epub 2019 Sep 12. PMID 31521672
- [Derived] Dunican EM, Elicker BM, Gierada DS, Nagle SK, Schiebler ML, Newell JD, Raymond WW, Lachowicz-Scroggins ME, Di Maio S, Hoffman EA, Castro M, Fain SB, Jarjour NN, Israel E, Levy BD, Erzurum SC, Wenzel SE, Meyers DA, Bleecker ER, Phillips BR, Mauger DT, Gordon ED, Woodruff PG, Peters MC, Fahy JV; National Heart Lung and Blood Institute (NHLBI) Severe Asthma Research Program (SARP). Mucus plugs in patients with asthma linked to eosinophilia and airflow obstruction. J Clin Invest. 2018 Mar 1;128(3):997-1009. doi: 10.1172/JCI95693. Epub 2018 Feb 5. PMID 29400693
- See also: Severe Asthma Research Program Main Clinicaltrials.gov Webpage — http://www.clinicaltrials.gov/ct2/show/study/NCT01606826?term=severe+asthma+research+program&rank=1